CLINICAL TRIAL: NCT01059929
Title: A Double-blinded Randomized Controlled Trial of Dexmedetomidine Versus Propofol for Sedation in Mechanically Ventilated Medical Intensive Care Unit Patients.
Brief Title: Dexmedetomidine Versus Propofol in the Medical Intensive Care Unit (MICU)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: drug and placebo unavailable
Sponsor: University of Chicago (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16865B
Record Dates: First submitted 2009-09-14; First posted 2010-02-01 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Mechanical Ventilation; Critical Illness
Keywords: Hypnotics and Sedatives; Respiration, Artificial; Ventilators, Mechanical; Critical care; Intensive care; Physical therapy; Occupational therapy; Sedative medications
MeSH Terms: conditions — Critical Illness; Respiratory Aspiration | interventions — Dexmedetomidine; Propofol; Fentanyl; Midazolam; Restraint, Physical; Occupational Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Active Comparator): Patients in this arm will receive continuous dexmedetomidine infusion (0.2 - 1.5 mcg/kg/hour) titrated to the target Richmond Agitation Sedation Scale for the duration of mechanical ventilation or 7 days on study, whichever is first.
  Interventions: Drug: Dexmedetomidine; Drug: Fentanyl; Drug: Midazolam; Behavioral: Physical and Occupational Therapy
- Propofol (Active Comparator): Patients in this arm will receive propofol (5 - 50 mcg/kg/min) for sedation, titrated to the target Richmond Agitation Sedation Scale for the duration of mechanical ventilation or 7 days on study, whichever is first.
  Interventions: Drug: Propofol; Drug: Fentanyl; Drug: Midazolam; Behavioral: Physical and Occupational Therapy

INTERVENTIONS:
Drug: Dexmedetomidine — continuous IV infusion 0.2 - 1.5 ucg/kg/hour titrated to target RASS
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Propofol — continuous IV infusion (5 - 50 ucg/kg/min) titrated to target RASS
  Other Names: Diprivan
  Arms: Propofol
Drug: Fentanyl — 25 - 200 mcg IV every hour (as multiple IV pushes) as needed titrated to Non-Verbal Pain Scale
Drug: Midazolam — 0.01 - 0.1 mg/kg IV push every 10 minutes as needed for agitation (RASS>+2)
  Other Names: Versed
Behavioral: Physical and Occupational Therapy — Daily therapy sessions targeting range of motion, strength, and mobility

SUMMARY:
This is a randomized controlled trial to compare propofol to dexmedetomidine for prolonged sedation (> 24 hours) in critically ill patients who require mechanical ventilation.

DETAILED DESCRIPTION:
Mechanically ventilated critically ill patients are routinely given sedative and analgesic medications to relieve pain and anxiety associated with intubation, mechanical ventilation, and critical care in general. While integral in minimizing discomfort, these medications may increase mechanical ventilation time, the duration of intensive care unit (ICU) stay, ICU complications (e.g. delirium, ventilator associated pneumonia, venous thromboembolism), the morbidity associated with critical illness, and patient mortality. This study compares two sedative medications that have been used in patients who require a mechanical ventilator. Enrolled patients will be randomly assigned to receive propofol or dexmedetomidine for sedation while they require ventilatory support. All patients will also receive the pain medication fentanyl as needed.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* mechanically ventilated through endotracheal tube
* anticipated need for ventilation > 48 hours
* requiring sedative/analgesic medication

Exclusion Criteria:

* on mechanical ventilator > 96 hours
* primary neurologic disease
* post cardiac arrest
* do not speak English (assessment only English language validated)
* pregnancy or lactation
* active myocardial ischemia
* second or third degree heart block
* pancreatitis
* elevated serum triglycerides (> 400 mg/dL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Kress, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexmedetomidine | Propofol
Started | 20 | 21
Completed | 20 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine | Propofol | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Mean (Full Range); unit: years] | 60.5 [33 to 87] | 67 [21 to 89] | 63.8 [21 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 9 | 12 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 11 | 19
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Days With Delirium
Description: delirium assessment using CAM-ICU
Time Frame: daily up to 28 days
Population: Study terminated early due to inability to maintain study drug supply in investigational pharmacy.
Measure: Median (Inter-Quartile Range); unit: proportion of days
Arm/Group | Dexmedetomidine | Propofol
Number analyzed (Participants) | 20 | 21
proportion of days | 0 [0 to 0.71] | .33 [0.13 to 0.71]

2. Secondary Outcome: Drug Efficacy According to Richmond Agitation Sedation Scale (RASS) Score
Description: Richmond Agitation Sedation Scale (RASS). This is a validated scale that measures level of sedation. The scale ranges from -5 to +4. -5 refers to a state where one is unarousable, +4 refers to a state where one is combative. The median and inter-quartile range over all daily assessments will be provided.
Time Frame: Daily up to day 28
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dexmedetomidine | Propofol
Number analyzed (Participants) | 20 | 21
score on a scale | -1 [-1 to -0.57] | -1.6 [-3.23 to -1]

3. Secondary Outcome: Number of Patients Completing Mobility Milestones
Description: Milestones: sitting upright independently, standing independently, transfer to chair, marching in place, ambulating independently
Time Frame: Daily through day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine | Propofol
Number analyzed (Participants) | 20 | 21
Participants | 7 | 6

4. Secondary Outcome: Days on Ventilator
Time Frame: 60 days from enrollment
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Dexmedetomidine | Propofol
Number analyzed (Participants) | 20 | 21
days | 3.85 [2.28 to 16.6] | 4.05 [2.54 to 11.49]

5. Secondary Outcome: Days in ICU
Time Frame: 60 days from enollment
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Dexmedetomidine | Propofol
Number analyzed (Participants) | 20 | 21
days | 6.39 [3.64 to 17.6] | 5.61 [2.88 to 11.22]

6. Secondary Outcome: Mortality
Time Frame: 28 days from enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine | Propofol
Number analyzed (Participants) | 20 | 21
Participants | 8 | 12

7. Secondary Outcome: Number of Participants With ICU Complications
Time Frame: daily through day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine | Propofol
Number analyzed (Participants) | 20 | 21
Participants | 0 | 0

8. Secondary Outcome: Number of Patients Requiring Fentanyl
Time Frame: during infusion of study medication up to day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine | Propofol
Number analyzed (Participants) | 20 | 21
Participants | 3 | 6

9. Secondary Outcome: Number of Patients Requiring Midazolam
Time Frame: during infusion of study medication through day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine | Propofol
Number analyzed (Participants) | 20 | 21
Participants | 3 | 0

10. Secondary Outcome: Days in Hospital
Time Frame: 60 days from enrollment
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Dexmedetomidine | Propofol
Number analyzed (Participants) | 20 | 21
days | 14.33 [6.3 to 32.39] | 12.96 [4.83 to 20.82]

11. Secondary Outcome: Number of Patients Completing Activities of Daily Living
Description: activities of daily living: eating, bathing, dressing, grooming, toileting
Time Frame: daily through day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine | Propofol
Number analyzed (Participants) | 20 | 21
Participants | 7 | 6

12. Secondary Outcome: Number of Adverse Medication Effects
Time Frame: duration of infusion of study medication up to 28 days
Measure: Number; unit: number of events
Arm/Group | Dexmedetomidine | Propofol
Number analyzed (Participants) | 20 | 21
number of events | 0 | 0

ADVERSE EVENTS:
Arm/Group | Dexmedetomidine | Propofol
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No